CLINICAL TRIAL: NCT02061644
Title: Intraocular Pressure Changes After Spinal Anesthesia: Acute and Subacute Effects
Brief Title: Spinal Anesthesia - Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Dr. Ruslan Abdullayev, Adiyaman University Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Spinal-IOP
Record Dates: First submitted 2014-02-10; First posted 2014-02-13 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Intraocular Pressure
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal (Experimental): Spinal anesthesia for surgical procedure will be applied to the patients. Intraocular pressures will be measured before and after the procedure.
  Interventions: Other: Spinal anesthesia

INTERVENTIONS:
Other: Spinal anesthesia — Routine spinal anesthesia procedure will be made to the patients for surgical anesthesia.

SUMMARY:
We aim to investigate the effect of spinal anesthesia on intraocular pressure.

DETAILED DESCRIPTION:
Spinal anesthesia provides adequate anesthetic conditions for many operations. These operations include orthopedic, urological, gynecological and many general surgery operations. Although few, side effects of the procedure and its effects on body are well known. However, there is inadequate knowledge about the effects of spinal anesthesia on pressure changes in the eyes. These pressure changes in eyes can result in some detriments. Elevated pressures in the eyes can result in disease known as glaucoma, that makes hazard to eyes. Decreased eye pressures can also result in some eye detriments.

We aimed to investigate the effects of spinal anesthesia procedure on eye (intraocular) pressure changes.

ELIGIBILITY:
Inclusion Criteria:

* patients having general surgery operations under umbilicus
* patients of American Society of Anesthesiologists (ASA) status I-II

Exclusion Criteria:

* patients denying spinal anesthesia
* contraindications for spinal anesthesia
* eye diseases
* hypertension
* ASA status III or more

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of the patients with changed intraocular pressure | One month

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Dr, Principal Investigator — Adiyaman University Research Hospital, Department of Anesthesiology and Reanimation, Adiyaman City, Turkey.
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Turkey (Türkiye)